CLINICAL TRIAL: NCT01033305
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study of a Controlled Release Minicapsule Formulation of Ciclosporin (CyCol™) in the Treatment of Mild to Moderate Ulcerative Colitis
Brief Title: Oral Ciclosporin for Colonic Release in Ulcerative Colitis (CyCol™)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sigmoid Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYC-201
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Mild to Moderate Ulcerative Colitis
Keywords: UC
MeSH Terms: interventions — Cyclosporine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CyCol™ (Experimental)
  Interventions: Drug: CyCol™

INTERVENTIONS:
Drug: CyCol™ — Orally, once per day for 4 weeks
  Other Names: Ciclosporin
  Arms: CyCol™
Drug: Placebo — Orally, once per day for 4 weeks
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This is a multi-center study in Ireland and United Kingdom to determine the effects, safety and tolerability of a drug called CyCol™ in improving mild to moderate ulcerative colitis (UC).

Informed consent will be obtained and following confirmation of eligibility and disease assessment, study participants will be randomised (allocated by chance) to take either CyCol™, or placebo, orally once every day for four weeks. Study visit assessments will include blood and stool tests, physical examinations and flexible sigmoidoscopies (inspection of the bowel wall using a flexible camera).

Half the participants will receive CyCol™ and half will receive placebo. At the end of treatment (4 weeks) study participants will be reassessed again and the findings in those who received CyCol™ will be compared with those who received placebo. Any side effects experienced during the study and the safety of treatment with CyCol™ will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged > 18 years
* Diagnosis of mild to moderate diagnosis of UC involving at least the rectum and sigmoid colon
* Clinical severity assessed at screening using the Disease Activity Index (DAI)
* Clinical severity documented and confirmed by flexible sigmoidoscopy, within 7 days of starting study treatment
* Signed and dated written informed consent.
* Willing to maintain current UC medication dosing regimen from screening until the end of the 4-week treatment period.
* Able and willing to refrain from intake of St. Johns Wort or any other prescription, over-the-counter, or herbal preparation that is known to affect cytochrome P450 metabolism throughout the 4-week treatment period.
* Able and willing to refrain from intake of grapefruit or grapefruit juice or any other food or drink that is known to affect cytochrome P450 metabolism throughout the 4 week treatment period of the study.

Exclusion Criteria:

* Severe or fulminant UC.
* UC limited to rectum only.
* Any previous colonic surgery.
* Any histological evidence of dysplasia on colonoscopic biopsy.
* Women of childbearing potential who are unable or unwilling to use adequate contraceptive methods to avoid pregnancy.
* Previous unsuccessful ciclosporin therapy.
* Biologic therapy within the past 2 months prior to study treatment.
* Methotrexate therapy within 4 weeks of study treatment.
* A steroid treatment dose of greater than 10 mg/day prednisolone (or equivalent) within 4 weeks of study treatment.
* Use of topical treatment (e.g. enemas) within 4 weeks of study treatment and unwilling to refrain from use of topical treatments from the screening visit until the end of the 4-week treatment period.
* Significant renal impairment, hepatic impairment, uncontrolled hypertension, premalignant skin lesions or current malignancies, or any other severe co-morbid condition.
* Known hypersensitivity to ciclosporin or any of its excipients.
* Positive screening stool assay for Clostridium difficile, hemorrhagic E.coli 0157:H7, Salmonella or Shigella
* Diagnosis of Crohn's colitis, ischemic colitis, NSAID-induced colitis, or radiation colitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of CyCol™ in inducing clinical remission of mild to moderate Ulcerative Colitis. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diarmuid O'Donoghue, Prof, Principal Investigator — St Vincent's University Hospital, Ireland; Stuart Bloom, M.D., Principal Investigator — University College Hospital NHS Trust
Locations (22):
- Ireland (8):
  - Cork University Hospital, Cork, Co. Cork
  - Mater Misercordiae University Hospital, Dublin, Co. Dublin
  - St. James's Hospital, Dublin, Co. Dublin
  - Clinical Science Institute, Galway, Co. Galway
  - The Adelaide and The Meath Hospital (Tallaght), Tallaght, Dublin
  - Beaumont Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - MidWestern Regional Hospital, Limerick
- United Kingdom (14):
  - University College Hospital London, London, London
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell and West MidlandsHospitals NHS Trust, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Conventry university Hospital, Coventry
  - Leeds General infirmary, Leeds
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool
  - Kings College London, London
  - St. Mark's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - George Elliot hospital, Nuneaton
  - John Radcliff Hospital, Oxford
  - Royal Shrewsbury Hospital, Shrewsbury
  - New Cross Hospital, Wolverhampton

REFERENCES:
- See also: company website — http://www.sigmoidpharma.com